CLINICAL TRIAL: NCT04695808
Title: The Effect of Yoga Training on Menopausal Symptoms on Menopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Arzu Abiç, Senior İnstructor, Eastern Mediterranean University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Supportive Care
Other Study IDs: g9987n5g; Duygu Yılmaz Vefikulucay (Other: Eastern Mediterranean University)
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Menopause
Keywords: menopause; yoga; symptoms
MeSH Terms: interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Yoga practice will be done two days a week for 10 weeks.
  Interventions: Behavioral: yoga
- control group (No Intervention): no intervention

INTERVENTIONS:
Behavioral: yoga — Yoga practice will be done two days a week for 10 weeks.
  Arms: intervention group

SUMMARY:
Parallel to the increase in life expectancy by years, the population of women living in the post-menopausal period is also increasing. In order to have a healthy menopause, which is an important part of women's life, it is thought that the adoption of yoga practice without health risks by women and its implementation as a lifestyle may be effective in reducing the symptoms of menopause experienced by women. In line with this information, it is aimed to determine the effect of yoga training on menopausal symptoms. The research will be carried out with menopausal women between the ages of 40-60 in Famagusta region. Women will be divided into two groups as intervention and control. Personal information form and menopause rating scale will be used in the research. The intervention group will be given yoga practice two days a week for 10 weeks. Menopause rating scale will be applied to the intervention and control group before and after the research.

DETAILED DESCRIPTION:
Parallel to the increase in life expectancy by years, the population of women living in the post-menopausal period is also increasing. In order to have a healthy menopause, which is an important part of women's life, it is thought that the adoption of yoga practice without health risks by women and its implementation as a lifestyle may be effective in reducing the symptoms of menopause experienced by women. In line with this information, it is aimed to determine the effect of yoga training on menopausal symptoms. The research will be carried out with menopausal women between the ages of 40-60 in Famagusta region. Women will be divided into two groups as intervention and control. Personal information form and menopause rating scale will be used in the research. The intervention group will be given yoga practice two days a week for 10 weeks. Menopause rating scale will be applied to the intervention and control group before and after the research.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in research,
* Can read and write in Turkish,
* Open to communication,
* Those who are between the ages of 40-60 and do not experience menstruation for at least one year, Do not use medication to treat menopausal symptoms,
* No diagnosed musculoskeletal disease, no severe heart disease,
* Not doing regular exercise and yoga,
* Not surgically menopausal,
* Women without psychiatric problems

Exclusion Criteria:

* Refusing to participate in research,
* Can't read and write Turkish,
* Communication is not possible,
* Those who are younger than 40 or older than 60 have experienced menstruation for at least one year
* Using medication for the treatment of menopausal symptoms,
* Those with a diagnosed musculoskeletal disease, severe heart disease,
* Doing regular exercise and yoga,
* Surgically menopausal, Women with psychiatric problems

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women aged 40-60 who are in menopause
Enrollment: 62 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-11-29 (Actual)

PRIMARY OUTCOMES:
menopause rating scale | 3 months
  It was developed in German by Schneider et al. In 1992 to measure the severity of menopausal symptoms and was adapted to English in 1996. MRT was adapted to Turkish by Gürkan in our country in 2005. There are "0 = None", "1 = Mild", "2 = Moderate", "3 = Severe" and "4 = Very severe" options for each item in the Likert-type scale consisting of 11 items including menopausal complaints. The total score of the scale is calculated based on the scores given for each item. The lowest score that can be obtained from the scale is 0, the highest score is 44.

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern Mediterranean University, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Efficacy of yoga for vasomotor symptoms: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/24045673/
- See also: Efficacy of omega-3 for vasomotor symptoms treatment: a randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/23982113/
- See also: Hatha Yoga practice decreases menopause symptoms and improves quality of life: A randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/27261993/
- See also: Effects of Yoga and Aerobic Exercise on Actigraphic Sleep Parameters in Menopausal Women with Hot Flashes — https://pubmed.ncbi.nlm.nih.gov/27707450/